CLINICAL TRIAL: NCT07337031
Title: A Randomized Controlled Trial of Complex Behavioral Intervention on Prognostic Survival in Comprehensive Treatment of Patients With Unresectable Liver Cancer
Brief Title: A Trial of Behavioral Intervention on Prognostic Survival of Patients With Unresectable Liver Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, Luo Susu, Associate Professor, Eastern Hepatobiliary Surgery Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 25ZR1402578
Record Dates: First submitted 2025-12-17; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Primary Hepatocellular Carcinoma; Unresectable Liver Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- complex intervention group (Experimental)
  Interventions: Behavioral: complex behavioral intervention
- routine care group (No Intervention)

INTERVENTIONS:
Behavioral: complex behavioral intervention — Including behavioral intervention measures such as alcohol cessation management, smoking cessation and respiratory function training, nutrition management, exercise management, blood sugar and weight management, sleep management, pain management, wound and infection management, mindfulness meditation and mental health management.
  Arms: complex intervention group

SUMMARY:
Research purpose

1. To evaluate the impact of complex behavioral intervention on the one-year overall survival rate of patients with unresectable liver cancer after comprehensive treatment, a comparative study was conducted between the complex behavioral intervention group and the standard medical care control group, and the dose-response relationship between the intervention intensity and clinical outcomes was explored.
2. Analyze the impact mechanisms of complex behavioral interventions on patients' quality of life, adverse treatment reactions, and key biological indicators, including evaluating clinical outcomes such as 2-year overall survival rate, progression-free survival (PFS), objective response rate (ORR), and disease control rate (DCR), as well as the association between changes in related biomarkers and behavioral compliance.
3. Evaluate the implementation effect and sustainability of the "in-hospital face-to-face + wechat platform" hybrid intervention model, including intervention acceptance, long-term behavior maintenance, health economic benefits, and perioperative recovery of patients undergoing down-conversion surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically or radiologically confirmed primary hepatocellular carcinoma;
2. BCLC stage B-C, initially assessed as unresectable;
3. Age 18-75 years;
4. ECOG performance status score 0-2;
5. Child-Pugh classification grade A or B (<=9 points);
6. Normal cognitive ability, capable of understanding and following intervention protocols;
7. Both the patient and primary caregiver can use a smartphone and the WeChat platform and are able to complete questionnaires and follow-up tasks;
8. Voluntarily participates in the study and signs the informed consent form.

Exclusion Criteria:

1. Presence of malignant tumors in other organs;
2. Presence of extrahepatic metastasis;
3. Presence of any of the following severe organic diseases in any organ:

(1) Cardiovascular: NYHA class III-IV heart failure, acute coronary syndrome within the past 6 months; (2) Liver: Child-Pugh class C cirrhosis, or ALT/AST >5 times the upper limit of normal; (3) Kidney: eGFR <45 mL/min/1.73m^2 or dialysis-dependent; (4) Respiratory: respiratory failure requiring long-term oxygen therapy; (5) Hematologic: hemoglobin <9 g/dL or platelets <75×10^9/L; 4. History of psychiatric disorders, severe cognitive impairment, or substance abuse; 5. Previous liver transplantation or treatment for malignant liver tumors; 6. Complete thrombosis of the main portal vein; 7. Female patients who are pregnant or breastfeeding; 8. Presence of severe congenital or acquired immunodeficiency; 9. Unwillingness to sign the informed consent form; 10. Other conditions deemed unsuitable for participation in this study by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival rate | The time from enrollment to death caused by any reason, mainly the one-year survival rate

SECONDARY OUTCOMES:
2-year overall survival rate | The survival rate from enrollment to two years after intervention
Progression-Free Survival | The time from enrollment to disease progression (according to the mRECIST 2010 version) or death caused by any reason, assessed up to 36 months (this study will last for 36 months)
Disease-Free Survival | From the date of surgery to disease recurrence, progression, or death due to any cause, whichever occurs first, assessed up to 36 months (this study will last for 36 months)
Objective Response Rate | assessed up to 36 months (this study will last for 36 months)
  The proportion of patients achieving complete remission (CR) or partial remission (PR) (according to the mRECIST 2010 version)
Disease Control Rate | assessed up to 36 months (this study will last for 36 months)
  The proportion of patients achieving complete response (CR), partial response (PR), or stable disease (SD) (according to the mRECIST 2010 version)
Treatment-related adverse reactions | assessed up to 36 months (this study will last for 36 months)
  From the moment of enrollment. Collected using the PRO-CTCAE (Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events) scale.
HCC Quality of life | assessed up to 36 months (this study will last for 36 months)
  Collected using the EORTC QLQ-L13 scale

CONTACTS AND LOCATIONS:
Locations (1):
- Eastern Hepatobiliary Surgery Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No